CLINICAL TRIAL: NCT00318825
Title: Use of Nitrous Oxide for Analgesia During Colonoscopy - A Randomised Trial
Brief Title: Nitrous Oxide for Analgesia During Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rikshospitalet University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: s-05225
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2006-04

CONDITIONS: Pain
Keywords: Pain; Colonoscopy; Sedation
MeSH Terms: conditions — Pain | interventions — Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous oxide

SUMMARY:
The purpose of the study is to determine the analgetic effect of nitrous oxide during colonoscopy, compared to no sedation and intravenous (IV) sedation.

DETAILED DESCRIPTION:
Background

Colonoscopy is the gold standard for diagnosis and endoscopic treatment of diseases in the colon and rectum (1). However, many patients experience discomfort during the procedure. Therefore, IV sedation and/or analgesia is routinely given during colonoscopy at the majority of centers around the world.

Midazolam, the most frequent sedative, is a benzodiazepine with hypnotic and sedative effects (2). The half-life of the substance is about 1-2.5 hours, and thus substantially longer than the duration of a colonoscopy (approximately 30 minutes). Additionally, Midazolam gives pronounced amnesia that lasts even longer than the hypnotic effect. Opioids are also frequently used during colonoscopy, with Pethidine as the most common one (half-life: 3 hours).

Use of the above mentioned drugs make it necessary to closely monitor the patients after colonoscopy for several hours, often in specially designed resource-demanding recovery units. Furthermore, due to the amnesia, it is often not possible to give information about findings and further work-up or surveillance to patients after colonoscopy. Finally, patients are not allowed to drive a car for the rest of the day after IV sedation during colonoscopy (2).

Nitrous oxide (N2O) is used as an inhalative gas during anesthesia, labour and at some dentist practices, most frequent in a fixed 50:50 combination with O2. N2O has a strong analgetic effect, and none or only slight sedative effects in concentrations < 80%. N2O has a very rapid onset of effect (a few seconds), and its half-life in the human body after the stop of inhalation is shorter than 1 minute (3). Patients receiving N2O in a 50:50 combination with O2 are awake, don't need post-procedure recovery and may drive their own car home (4). However, as N2O diffuses quickly through biological membranes, caution is warranted when used for patients with the following conditions: sinusitis, otitis, ileus, bowl obstruction, and megacolon. Pregnant women should not be exposed to N2O.

There are some small studies showing good analgetic effects of N2O during colonoscopy, without significant side-effects (5,6,7). One additional study, however, reported on the poor effects of N2O during colonoscopy (8). This study has, however, been subject for critique because it lacks in methodology (9).

N2O is currently used only at some hospitals around the world.

The use of N2O in colonoscopy instead of IV drugs seems to be attractive for several reasons:

* Adequate analgesia without disturbing sedation during the procedure. The patient is awake and co-operative.
* No amnesia. All information can be given to the patient immediately after the procedure.
* The patient can control inhalation of the analgetic N2O himself. This may enhance patient satisfaction.
* Rapid stop of effect after stopped administration. No surveillance needed, patients can leave the hospital immediately.
* N2O does not impair psychomotoric abilities (4,10). Thus, patients may use their own car to and from the appointment. This is resource-sparing for the patient and/or payer. Moreover, it may increase compliance for colonoscopy in rural areas.

Hypothesis/endpoint

Primary endpoint:

* Does the use of N2O during colonoscopy result in adequate analgesia for the patient?

Secondary endpoints

* Are there any side-effects due to the use of N2O during colonoscopy?
* Is there a reduction in the number of patients needing IV sedation?
* Is there any dose reduction of IV drugs?

Methods

The study is a randomised, controlled, double-blinded, single-center trial. Participants, after giving written informed consent, are randomised to one of two treatment groups:

1. Group 1: N2O inhalation (verum)
2. Group 2: O2 inhalation (placebo)

All patients in both groups will start their examination without any use of sedatives/analgetics. On demand, the patients will then be instructed to use the mask for inhalation of gas (N2O in verum group, O2 in placebo group). In case of insufficient effect of inhalation, patients in both groups will be given midazolam and/or pethidine until satisfactorily relieved from pain or discomfort.

Both the patient and the endoscopist are blinded with regard to the type of gas used. The endoscopy assistant handles the gas couplings on scene. Randomisation will be done 1:1 for the groups, in blocks of 6 patients, using a computer program and sealed envelopes for concealment on scene.

Study medication

N2O or O2 is to be administrated by inhalation via a mouth/nose mask. N2O and O2 is delivered by the central hospital gas system. The mask contains a tight circle, where gas is only released from the mask by negative pressure from inspiration of the patient. This is to prevent leakage of gas to the environment. The mask is held by the patient and the patient controls the use of the mask (patient-controlled analgesia). The gas system has been approved by the local department of medical equipment. Measurements of N2O concentrations in the endoscopy room are frequently performed by an independent body, in accordance with Norwegian law.

Midazolam (standard dose 2.5 mg) and pethidin (standard dose 25 mg) are used as IV drugs.

Stopping rules

If any adverse effects are observed, blinding is to be broken. The endoscopist decides changes in the sedation procedure, as appropriate in the individual situation.

Measurement of pain and discomfort

After the examination, study participants receive a questionnaire about pain and discomfort during and after the examination. This questionnaire has been used in our department for several years, and is validated for the use in colonoscopy (11, 12). The questionnaire contains a 4-point scale (4-VRS) for the patient's characterisation of pain and discomfort. Additionally, the questionnaire asks about any side-effects observed by the patient.

The questionnaire is to be filled in by the patient at home the day after the procedure, and to be mailed back to the center in a prepaid envelope.

Exclusion criteria:

1. Patients who don't understand information given
2. Age under 18 years
3. Pregnancy
4. Otitis/sinusitis
5. Ileus/bowel obstruction
6. Megacolon
7. Suspected pneumothorax

Power calculation

As there is only limited knowledge from the literature, we will perform a pilot study including 10 patients in each group. The data of the pilot study will then serve for a power calculation to find out the number of individuals needed in the study.

Ethics

The Norwegian version of the protocol has been approved by the regional ethics committee of Southern Norway (no. S-05225). The Norwegian Data Inspectorate has been informed about the study (no. 25660). The study is registered in a clinical trials registry (www.clinicaltrials.gov).

Ownership and publication

All generated data are owned by Rikshospitalet University Hospital. A manuscript dealing with the data will be submitted to a medical journal for publication, regardless of the nature of the results. Authorship will be according to the Vancouver rules (13).

Literature

1. Aabakken L. Gastrointestinal endoskopi. Oslo 1997
2. Felleskatalogen 2004. Felleskatalogen as, Oslo 2004
3. Forth W, et al. Pharmakologie und Toxikologie. Wissenschaftsverlag. Mannheim 1992
4. Martin JP, et al. Inhaled patient-administered nitrous oxide/oxygen mixture does not impair driving ability when using as analgesia during screening flexible sigmoidoscopy. Gastrointest Endosc 2000;51:701-3.
5. Harding TA, et al. The use of inhaled nitrous oxide for flexible sigmoidoscopy: a placebo-controlled trial. Endoscopy 2000;32:457-80
6. Notini-Gudmarson AK, et al. Nitrous oxide: a valuable alternative for pain relief and sedation during routine colonoscopy Endoscopy 1996;28:283-7
7. Hedenbro J, et al. Lustgas øverlæget vid koloskopi. Lakartidningen 1996;93:257-8
8. Forbes GM, Collins BJ. Nitrous oxide for colonoscopy; a randomized controlled study. Gastrointest Endosc 2000;51:271-7.
9. Faddy SC. Substantial surveillance bias in an unblended study of pain and adverse effects associated with nitrous oxide inhalation or standard medication for colonoscopy. Gastrointest Endosc 2001;54 (letter).
10. Trojan J, et al. Immediate recovery of psychomotor function after patient-administered nitrous oxide/oxygen inhalation for colonoscopy. Endoscopy 1997;29:17-22
11. Bretthauer M, et al. A randomized controlled trial to assess the safety and efficacy of carbon dioxide insufflation in colonoscopy. Gut 2002;50:604-7
12. Skovlund E, et al. Sensitivity of pain rating scales in an endoscopy trial. J Clin Pain, 2005, in press
13. Uniform requirements for manuscripts submitted to biomedical journals: writing and editing for biomedical

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for colonoscopy

Exclusion Criteria:

* Patients who don't understand information given
* Age under 18 years
* Pregnancy
* Otitis/sinusitis
* Ileus/bowel obstruction
* Megacolon
* Suspected pneumothorax

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Does the use of nitrous oxide (N2O) during colonoscopy result in adequate analgesia for the patient?

SECONDARY OUTCOMES:
Are there any side-effects due to the use of N2O during colonoscopy?
Is there a reduction in the number of patients needing IV sedation?
Is there any dose reduction of IV drugs?

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bretthauer, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Loberg M, Furholm S, Hoff I, Aabakken L, Hoff G, Bretthauer M. Nitrous oxide for analgesia in colonoscopy without sedation. Gastrointest Endosc. 2011 Dec;74(6):1347-53. doi: 10.1016/j.gie.2011.07.071. PMID 22136779